CLINICAL TRIAL: NCT06997562
Title: Comparative Efficacy of Greater Occipital Nerve Blockade and Sphenopalatine Ganglion Blockade in Patients With Episodic Migraine
Brief Title: Greater Occipital Nerve Blockade and Sphenopalatine Ganglion Blockade in Patients With Episodic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Omar Twaisy, Lecturer of Anesthesia and Intensive Care, Faculty of Medicine, New Valley University, Egypt., New Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250430007
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Greater Occipital Nerve Block; Sphenopalatine Ganglion Block; Episodic Migraine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Greater occipital nerve blockade group (Experimental): Patients will receive greater occipital nerve blockade using 2 mL of 2% lidocaine at the medial one-third of the line between the occipital protuberance and mastoid process.
  Interventions: Other: Greater occipital nerve blockade
- Sphenopalatine ganglion blockade group (Experimental): Patients will receive greater sphenopalatine ganglion blockade using 2 mL of 2% lidocaine using a transnasal approach with a cotton swab inserted along the superior middle turbinate to the posterior nasopharyngeal wall.
  Interventions: Other: Sphenopalatine ganglion blockade

INTERVENTIONS:
Other: Greater occipital nerve blockade — Patients will receive greater occipital nerve blockade using 2 mL of 2% lidocaine at the medial one-third of the line between the occipital protuberance and mastoid process.
  Arms: Greater occipital nerve blockade group
Other: Sphenopalatine ganglion blockade — Patients will receive greater sphenopalatine ganglion blockade using 2 mL of 2% lidocaine using a transnasal approach with a cotton swab inserted along the superior middle turbinate to the posterior nasopharyngeal wall.
  Arms: Sphenopalatine ganglion blockade group

SUMMARY:
This study compares the effectiveness of greater occipital nerve blockade and sphenopalatine ganglion blockade in reducing headache intensity, duration, frequency, and disability in patients with episodic migraine.

DETAILED DESCRIPTION:
Migraine is a chronic neurological disorder characterized by recurrent headaches, affecting millions globally. Peripheral nerve blocks such as Greater Occipital Nerve (GON) and Sphenopalatine Ganglion (SPG) blockade have emerged as promising non-pharmacologic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Both sexes.
* Diagnosed with episodic migraine per the International Classification of Headache Disorders, 3rd edition (ICHD-3).
* Failure to achieve adequate relief with at least one prophylactic migraine treatment.

Exclusion Criteria:

* Chronic migraine (≥15 headache days per month).
* History of nerve blocks within the last 6 months.
* Known allergy to anesthetic agents.
* Pregnancy or lactation.
* Active psychiatric conditions affecting compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-03 (Actual); Study Completion 2025-05-03 (Actual)

PRIMARY OUTCOMES:
Degree of headache intensity | 3 months post-procedure
  Reduction in headache intensity will be recorded using numeric rating scale (NRS). Each patient will be instructed about pain assessment with NRS score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable").

SECONDARY OUTCOMES:
Migraine disability assessment score | 3 months post-procedure
  The migraine disability assessment scores are as follows: little or no disability, 5 to 10; moderate disability, 1 to 20; and severe disability, more than 20.
Headache duration | 3 months post-procedure
  Headache duration will be recorded.
Headache frequency | 3 months post-procedure
  Headache frequency will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- New Valley University, New Valley, New Valley Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.